CLINICAL TRIAL: NCT05405738
Title: Effect of 2 Flap Palatoplasty Versus Furlow With Buccinators Flap During Palatal Cleft Repair on the Maxillary Development Patterns in Comparison to Non-cleft Children at 5-6years of Age
Brief Title: Cleft Palate Technique and Maxillary Growth
Status: Completed | Type: Observational
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohsen, principal investigator, Fayoum University
Other Study IDs: 2
Record Dates: First submitted 2022-05-22; First posted 2022-06-06 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Cleft Palate; Growth
MeSH Terms: conditions — Cleft Palate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- normal group
  Interventions: Other: normal group
- 2flap palatoplasty group
  Interventions: Procedure: 2 flap palatoplasty technique
- Furlow with buccinator group
  Interventions: Procedure: Furlow with buccinator technique

INTERVENTIONS:
Procedure: 2 flap palatoplasty technique — cleft palate repair by 2 flap palatoplasty technique
  Groups: 2flap palatoplasty group
Other: normal group — control normal group
  Groups: normal group
Procedure: Furlow with buccinator technique — cleft palate repair by Furlow with buccinator technique
  Groups: Furlow with buccinator group

SUMMARY:
comparison of the maxillary growth between cleft palate patients that underwent to repair by 2 flap palatoplasty versus Furlow with buccinator technique

ELIGIBILITY:
Inclusion Criteria:

* 5-6 years old childreen with previous treated complete cleft lip and palate, nonsyndromic.
* lip and palate repair performed by one craniofacial surgeon

Exclusion Criteria:

* Patients with syndromic cleft lip.
* Redu cases
* Bilateral cleft lip
* Patient older 6years or younger 5 years.
* Associated Cardiac anomalies.
* Any systemic condition

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 5-6ys old child with treated cleft palate
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2022-05-06 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
maxillar growth | through study completion, an average one week
  evaluation of the maxillary growth through Inter-canine width (ICW) measurement by mm

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum University, Al Fayyum, Egypt

REFERENCES:
- [Derived] Aboulhassan MA, Refahee SM, Sabry S, Abd-El-Ghafour M. Effects of two flap palatoplasty versus furlow palatoplasty with buccal myomucosal flap on maxillary arch dimensions in patients with cleft palate at the primary dentition stage: a cohort study. Clin Oral Investig. 2023 Sep;27(9):5605-5613. doi: 10.1007/s00784-023-05182-0. Epub 2023 Aug 2. PMID 37530892